CLINICAL TRIAL: NCT05697640
Title: A Parallel-group Treatment, Phase 2a, Double-blind, Placebo-controlled 2-arm Study to Show Improvement of Physical Function in SF-36 (SF-36-PF) in Participants Treated With Vericiguat Compared to Placebo Tablets in Male and Female Participants Aged 18-50 Years With Post-COVID-19 Syndrome Without (PCS) or With (PCS/CFS) Fulfillment of ME/CFS Criteria (VERI-LONG).
Brief Title: Study to Investigate Improvement in Physical Function in SF-36 With Vericiguat Compared With Placebo in Participants With Post-COVID-19 Syndrome
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Judith Bellmann-Strobl, Senior physician, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VERI-LONG; 01EP2201 (Other Grant/Funding Number: BMBF)
Record Dates: First submitted 2023-01-23; First posted 2023-01-26 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Post-COVID ME/CFS
Keywords: Post-COVID Syndrome; Long COVID; Chronic Fatigue Syndrome
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Fatigue Syndrome, Chronic | interventions — vericiguat

STUDY DESIGN:
Intervention Model Description: Two-arm parallel-group, randomized, placebo-controlled, double-blind, single-centre clinical trial in participants with post-COVID syndrome with and without ME/CFS.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vericiguat Oral Tablet (Active Comparator): Tested IMP: Vericiguat (film-coated tablet). Authorization status: Not authorised in this targeted therapeutic indication; Vericiguat is authorized for the dosages that will be administered in this trial for another indication. The tablets used in this trial are no trade product, but a special trial product produced and provided by the marketing authorization holder Bayer.
  Administration: Once daily (oral). Planned dosage: Three different dosages starting with 2.5 mg for two weeks, followed by 5 mg for two weeks and 10 mg for six weeks. The general IMP titration regimen was investigated and proven to be safe (max. dosages 10 mg/day) in patients with heart failure and reduced ejection fraction (Armstrong et al., 2020).
  Interventions: Drug: Vericiguat Oral Tablet
- Placebo Oral Tablet (Placebo Comparator): Comparator IMP: Placebo (film-coated tablet). Authorization status: Not authorised. The tablets used in this trial are no trade product, but a special trial product produced and provided by the marketing authorization holder Bayer.
  Administration: Once daily (oral). Planned dosage: Three different dosages starting with 2.5 mg for two weeks, followed by 5 mg for two weeks and 10 mg for six weeks to have identical conditions to verum.
  Interventions: Drug: Vericiguat Oral Tablet

INTERVENTIONS:
Drug: Vericiguat Oral Tablet — The treatment period includes ten weeks of daily vericiguat or placebo intake (depending on randomization) and a 30-day follow-up period (no vericiguat/placebo intake).

SUMMARY:
The goal of this clinical trial is to evaluate the therapeutic value of an approved drug (Vericiguat) in patients with post-COVID-19 syndrome, who suffer from profound tiredness or fatigue, regardless of bed rest.The main questions it aims to answer are: • Does Vericiguat relieve fatigue and/or other symptoms associated with post-COVID-19 syndrome? • What are the side effects of Vericiguat in this patient population; and how common are they?

Participants will be asked to participate for approx. 18 weeks. After screening, participants will receive assigned intervention of either 10 weeks of treatment with Vericiguat or matching placebo tablet, followed by 30 day follow-up period. Every participant will undergo trial, cardiovascular safety, and monitoring assessments.

The results of this study will provide information on whether Vericiguat can alleviate PCS-related symptoms as well as insights into the pathophysiological processes of PCS, which in turn can help to develop therapies.

DETAILED DESCRIPTION:
Although of high socioeconomic relevance, the pathomechanisms of post-COVID-19 syndrome (PCS) are not well understood and there is no established therapy. Preliminary evidence suggests that systemic tissue and organ hypoperfusion, resulting from impaired microvascular blood flow secondary to chronic endothelial dysfunction (ED), plays a key role in many symptoms.

The objective is to demonstrate improvement in physical function measured using the short form-36 health questionnaire (SF-36) in patients with post-COVID-19 syndrome with or without fulfillment of ME/CFS criteria treated with Vericiguat compared with placebo. Vericiguat is a drug that bridges endothelial dysfunction to improve microvascular perfusion and tissue and organ blood flow.

This is a two-arm parallel-group, randomized, placebo-controlled, double-blind, single-centre clinical trial in participants with PCS and PCS/CFS. Patients participate for approx. 18 weeks. Participants will be stratified according to diagnosis (with vs. without ME/CFS) and sex, and randomly assigned 1:1 after a screening phase of up to 28 days to receive assigned intervention of either 10 weeks of treatment with Vericiguat (including titration phase) or placebo, followed by 30 days follow-up period. One group receives a tablet of Vericiguat once daily for 10 weeks with a dosage titration to tolerated dose of 2.5 mg for 2 weeks, 5 mg for 2 weeks, 10 mg for 6 weeks. The other group receives a matching placebo tablet once daily for 10 weeks with the same titration regimen to ensure blinding. The starting dose is 2.5 mg Vericiguat or matching placebo, once daily, and a controlled and blood pressure-tolerated titration regimen will be used to achieve the anticipated target dose of 10 mg Vericiguat or matching placebo. Every participant will undergo trial, cardiovascular safety, and monitoring assessments. During the screening visit, the study team i) records the patient's medical history, ii) checks the in- and exclusion criteria, iii) performs a medical check-up, iv) performs an echocardiogram, and v) measures the patient's vital parameters. In female participants, a pregnancy test is carried out 5 times during the study.

The results of this study will provide information on whether Vericiguat can alleviate PCS-related symptoms such as fatigue, cognitive impairment, and impaired physical function (e.g., walking, stair climbing) and/or modulate paraclinical markers such as parameters of endothelial function. Moreover, the clinical trial will provide insights into the pathophysiological processes of PCS, which in turn can help to elucidate the disease etiology and to develop effective therapies.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adult who is 18-50 years old
* Confirmed (PCR or serology), non-hospitalized, mild to moderate acute COVID-19 cases according to WHO criteria with proven chronic ED and either: ME/CFS Canadian Consensus Criteria (CCC) with post exertional malaise (PEM) 2 - 14 hours = PCS or ME/CFS CCC criteria with PEM > 14 hours = PCS/CFS
* Ongoing symptoms of PCS or PCS/CFS for ≥ 6 months
* Bell Score: 30-60
* Evidence for endothelial dysfunction (ED) [as indicated by reactive hyperemia index (RHI) < 1.8 and/or ET-1 level > 90 percentile of healthy age- and gender matched controls or muscle fatigue (below cut-off values of area under the curve reference values for age-matched healthy controls and/or pathological optical coherence tomography angiography (OCTA))]
* For female subjects: Confirmed post-menopausal state (defined as amenorrhea for at least 12 months) or for women of childbearing potential: Negative highly sensitive urine or serum pregnancy test before inclusion/randomisation and practicing a highly effective birth control method (failure rate of less than 1 %):

  * combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral/intravaginal/transdermal), or
  * progestogen-only hormonal contraception associated with inhibition of ovulation (oral/injectable/implantable), or
  * intrauterine device, or
  * intrauterine hormone-releasing system, or
  * bilateral tubal occlusion, or
  * vasectomised partner, or
  * heterosexual abstinence.

Exclusion Criteria:

* COVID-19 vaccination within the last 4 weeks before inclusion
* Pre-COVID history of chronic fatigue syndrome or other fatigue syndromes that are due to associated diseases (e.g., cancer, autoimmune diseases [patients with a preexisting Hashimoto thyroiditis and/or fibromyalgia without fatigue syndromes can be included])
* Concomitant use of Vericiguat due to other diseases
* Contraindications against IMP
* Concurrent or anticipated concomitant use of PDE-5 inhibitors such as vardenafil, tadalafil, and sildenafil, nitrates, or sGC-stimulators
* Use of other sGC stimulators, e.g., riociguat
* Hypersensitivity to the active substance or any of the other ingredients
* Systolic blood pressure: < 100 mmHg at screening
* Known SARS-CoV-2 infection-related organ damage/comorbidity
* Severe renal or hepatic insufficiency
* Pregnancy or breastfeeding

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 104 (Estimated)
Dates: Start 2023-06-22 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Improvement in Physical Function (PF) as measured by the Short Form 36 Health Survey Questionnaire (SF-36) | 10 weeks after first IMP intake
  The Short Form 36 Health Survey (SF-36) is an established and widely used health-related quality of life measure. The Physical Function (PF) domain asks patients to report limitations on ten mobility activities, such as walking specified distances, carrying groceries, and bathing or dressing. Scores are weighted and transformed into a scale ranging from 0 (greatest possible health restrictions, i.e., severe disability) to 100 (no health restrictions). An intra-patient change of 10 points in SF-36-PF from baseline to week ten is considered clinically meaningful.

SECONDARY OUTCOMES:
Difference in responder rate in Physical Function (PF) as measured by the Short Form 36 Health Survey Questionnaire (SF-36) comparing Vericiguat with placebo | 10 weeks after first IMP intake
  Occurrence of responders in patients that receive Vericiguat compared with placebo. Responders are defined as an intra-patient 10-point increase in SF-36-PF from baseline to week ten.
Improvement in other sub-domains of the Short Form 36 Health Survey Questionnaire (SF-36) comparing Vericiguat with placebo | 10 weeks after first IMP intake
  Intra-patient change in other SF-36 subdomains from baseline to week ten.
Improvement in fatigue as measured by the Fatigue Severity Score (FSS) | 10 weeks after first IMP intake
  The Fatigue Severity Scale (FSS) is a 9-item scale that measures the severity of fatigue and its effect on a person's activities and lifestyle. Answers are scored on a seven-point scale (1 = strongly disagree; 7 = strongly agree). Thus, the minimum score is 9 (no fatigue), and the highest is 63 (heavy fatigue). Intra-patient change in fatigue severity from baseline to week 10 will be documented as indexed by the FSS.
Improvement in severity of muscle pain and headache as measured by the Canadian Consensus Criteria (CCC) symptom score | 10 weeks after first IMP intake
  The Canadian Consensus Criteria (CCC) Symptom Score quantifies ME/CFS symptoms. Its score ranges from 1 (no symptoms) to 10 (extreme symptoms). Intra-patient change in muscle pain and headache from baseline to week ten.
Improvement in symptoms of myalgic encephalomyelitis (ME)/ chronic fatigue syndrome (CFS) as measured by Canadian Consensus Criteria (CCC) Symptom Score | 10 weeks after first IMP intake
  Intra-patient change in ME/CFS symptoms from baseline to week 10 will be documented as indexed by the CCC Symptom Score.
Improvement in functional disability as measured by the Bell disability scale | 10 weeks after first IMP intake
  The Bell disability scale is a standard assessment in ME/CFS that evaluates functional ability in adult ME/CFS patients. Eleven statements describe patient status such as level of symptoms at rest, level of symptoms with exercise, activity level, and ability to perform work, travel and self care. Its score ranges from 0 (bedridden) to 100 (no symptoms). Intra-patient change in Bell score from baseline to week ten.
Improvement in symptoms of autonomic dysfunction as measured by the Composite Autonomic Symptom Score (COMPASS-31) | 10 weeks after first IMP intake
  The Composite Autonomic Symptom Score (COMPASS-31) is a refined, internally consistent, and markedly abbreviated quantitative measure of autonomic symptoms. It is based on the original Autonomic Symptom Profile (ASP) and COMPASS, applies a much-simplified scoring algorithm, and is suitable for widespread use in autonomic research and practice. It evaluates six domains of autonomic function: orthostatic intolerance, vasomotor, secretomotor, gastrointestinal, bladder, and pupillomotor domains. The score ranges from 0 (no symptoms) to 100 (strong autonomic dysfunction). Intra-patient change in autonomic dysfunction from baseline to week ten will be documented as indexed by the COMPASS-31.
Improvement in disease severity based on self- reported symptoms as measured by the Munich Berlin Symptom Questionnaire (MBSQ) | 10 weeks after first IMP intake
  The Munich Berlin Symptom Questionnaire (MBSQ) is a questionnaire for ME/CFS that captures the IOM and CCC diagnostic criteria as well as a total of 44 symptoms from 8 domains on a scale of 0 - 4 for frequency and severity. From this, a score for total symptom severity ranging from 0 (not present) to 352 (very severe) is calculated. Intra-patient change in MBSQ score from baseline to week ten.
Improvement in disease severity based on self- reported symptoms as measured by the Munich Long Covid Symptom Questionnaire (MLCSQ) | 10 weeks after first IMP intake
  The Munich Long Covid Symptom Questionnaire (MLCSQ) is a long covid questionnaire that measures a total of 83 symptoms from 13 domains on a scale of 1-3 for frequency and severity. This results in a score for total symptom severity ranging from 83 (mild) to 496 (severe). Intra-patient change in MLCSQ score from baseline to week ten.
Improvement in post exertional malaise (PEM) frequency, strength and severity as measured by the PEM questionnaire | 10 weeks after first IMP intake
  The PEM questionnaire determines frequency (from 0 to 20 points, higher scores equate to greater frequency), severity (from 0 to 20 points, higher scores equate to greater severity), and length (from 0 to 6 points, higher scores equate to longer duration) of PEM. Intra-patient change in PEM score from baseline to week ten.
Improvement in muscle fatigue measured by the repetitive hand grip strength test (HGS) | 10 weeks after first IMP intake
  Intra-patient change in hand grip strength (HGS) from baseline to week ten.
Improvement in orthostatic intolerance measured by the passive standing test | 10 weeks after first IMP intake
  Intra-patient change in blood pressure, sitting and standing heart rate, and delta heart rate from baseline to week ten.
Improvement of endothelial cell function as assessed using EndoPAT | 10 weeks after first IMP intake
  Intra-patient change in vascular regulation as indexed by the reactive hyperemia index (RHI) from baseline to week ten.
Improvement in cognitive function measured by the Symbol Digit Modalities Test (SDMT) | 10 weeks after first IMP intake
  The Symbol Digit Modalities Test (SDMT) is a screening instrument commonly used to assess neurological dysfunction. It detects cognitive impairment as well as changes in cognitive functioning over time and in response to treatment. The scores range between 0 and 110 (higher scores equate to greater cognitive functioning). Intra-patient change in cognitive score from baseline to week ten.
Improvement in ET-1 serum levels | 10 weeks after first IMP intake
  Intra-patient change in ET-1 level from baseline to week ten.
Difference of occurring AE and SAE comparing Vericiguat with placebo (IMP safety). | 10 weeks after first IMP intake
  Occurrence of IMP side and adverse effects, assessed with AE, SAE and SUSAR reports

CONTACTS AND LOCATIONS:
Overall Officials: Judith Bellmann-Strobl, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité - Universitätsmedizin Berlin, Berlin, State of Berlin, Germany

REFERENCES:
- [Background] Armstrong PW, Pieske B, Anstrom KJ, Ezekowitz J, Hernandez AF, Butler J, Lam CSP, Ponikowski P, Voors AA, Jia G, McNulty SE, Patel MJ, Roessig L, Koglin J, O'Connor CM; VICTORIA Study Group. Vericiguat in Patients with Heart Failure and Reduced Ejection Fraction. N Engl J Med. 2020 May 14;382(20):1883-1893. doi: 10.1056/NEJMoa1915928. Epub 2020 Mar 28. PMID 32222134